CLINICAL TRIAL: NCT01971892
Title: Non Invasive Ventilation After Abdominal Surgery in Postoperative Acute Respiratory Failure: a Multicenter Randomized Controlled Trial.
Brief Title: Non Invasive Ventilation in Abdominal Postoperative Period
Acronym: NIVAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9015
Record Dates: First submitted 2013-08-19; First posted 2013-10-29 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Surgery; Trauma to the Abdomen; Acute Respiratory Failure
Keywords: Abdominal surgery;; Postoperative complication;; Acute respiratory failure;; Hypoxemia;; Intubation;; Non-invasive ventilation
MeSH Terms: conditions — Abdominal Injuries; Postoperative Complications; Hypoxia | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non invasive ventilation (NIV) (Experimental): Experimental arm = non invasive ventilation (NIV) which associated pressure support ventilation (PSV: 5 to 15 cmH2O) and positive end expiratory pressure (PEEP: 5 to 10 cmH2O) NIV will intermittently delivered to the patients for at least six hours (cumulative tme of all trials which lasted at least 30 min) during the first 24h after the initiation of treatment. Between each NIV period, the patient will received supplemental oxygen through facial mask to achieve an oxygen saturation level above 94%.
  Interventions: Other: Non Invasive ventilation (facial mask and NIV ventilator)
- standard oxygen therapy with facial mask (Active Comparator): Patients assigned to standard medical therapy will received supplemental oxygen via a facial Venturi mask at a rate of up to 15 liters per minute with in order to maintain peripheral oxygen saturation above 94%.
  Interventions: Other: Standard oxygen therapy with facial mask

INTERVENTIONS:
Other: Non Invasive ventilation (facial mask and NIV ventilator) — Non invasive ventilation (NIV) which associated pressure support ventilation (PSV: 5 to 15 cmH2O) and positive end expiratory pressure (PEEP: 5 to 10 cmH2O). NIW will be delivered through a facial mask with either NIV ventilator or ICU ventilator with NIV option
  Arms: Non invasive ventilation (NIV)
Other: Standard oxygen therapy with facial mask — facial Venturi mask
  Arms: standard oxygen therapy with facial mask

SUMMARY:
Acute respiratory failure may occur early in the postoperative course, requiring endotracheal intubation and mechanical ventilation in selected patients, thus increasing morbidity and mortality and prolonging intensive care unit (ICU) and hospital stay.We will perform a multicenter, prospective, randomized clinical trial to compare the efficacy of non invasive ventilation (NIV) which associated pressure support ventilation (PSV: 5 to 15 cmH2O) and positive end expiratory pressure (PEEP: 5 to 10 cmH2O) with standard oxygen therapy in the treatment of postoperative acute respiratory failure. We also set out to examine the hypothesis that early application of NIV may prevent intubation and mechanical ventilation in patients who develop acute respiratory failure after abdominal surgery.

DETAILED DESCRIPTION:
The Non-Invasive Ventilation After Surgery (NIVAS) is an investigator-initiated, multi-center, stratified, two-arm parallel-group trial with a computer-generated allocation sequence and electronic system based randomization. The study protocol and statistical analysis plan were approved for all centers by a central Ethics Committee (France) according to French law.The NIVAS study is conducted in accordance with the declaration of Helsinki and was registered on August 2013.All centers have a long experience with NIV (more than 10 years of NIV use for ARF, and more than 5 years of NIV use for ARF following abdominal surgery). Randomization will stratified by department, age (less or more 60 years), site of surgery (upper or lower abdominal) and according to the presence or absence of postoperative epidural analgesia as this may influence outcomes. Treatment assignments will concealed from patients, research staff, the statistician, and the data monitoring and safety committee.

ELIGIBILITY:
Inclusion Criteria:

Eligibility :

* age of more than 18 years
* scheduled for elective or not elective abdominal surgery requiring laparotomy or laparoscopy and general anesthesia.

Inclusion :

* acute respiratory failure occurring within the seven days of the surgery procedure which is defined as presence and persistence for at least 30 min and at least one of the two followings: 1) a respiratory rate of more than 30 breaths per minute and 2) clinical signs suggestive of respiratory muscle fatigue, increased work of breathing, or both, such as use of respiratory accessory muscles, paradoxical motion of the abdomen, or retraction of intercostal spaces
* hypoxemia defined by a PaO2 lower than 60 mmHg in ambient air or lower than 80 mmHg under 15 liters O2 or an arterial O2 saturation by pulse-oximetry (SpO2) lower than 90% (PaO2/FiO2< 200 mmHg).

Exclusion Criteria:

* Emergency procedure surgery (operation that must be performed as soon as possible and no longer than 12 hours after inclusion in the study)
* previous recruitment into another trial.
* Cardiopulmonary arrest
* Glasgow coma scale <8
* Absence of airway protective gag reflex
* Upper airway obstruction
* Pregnancy.
* Patients who refuse to undergo endotracheal intubation, whatever the initial therapeutic approach
* Chronic home non invasive ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09-16 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary end point for the comparison between noninvasive ventilation (NIV) and standard oxygen therapy will be the tracheal intubation within 7 days after the initiation of treatment. | primary end point will be evaluated within 7 days after the initiation of treatment.
  Endotracheal intubation.

SECONDARY OUTCOMES:
Gas exchange after one to two hours after inclusion in the protocol | one to two hours after inclusion in the protocol
  Gas exchange will be obtain from arterial blood gases from an arterial line (radial or femoral). Judgement criteria for gas exchange will be oxygenation evaluated by PaO2/FiO2 ratio and PaCO2.
nosocomial infections within the 14 days and mortality | At D-14 that means 14 days after initiation of treatment
  * Pulmonary infection
  * Urinary infection
  * Catherter related infection
  * Bacteriemia and Mortality
length of ICU | From inclusion until the study until discharge or at 90 days maximal of ICU
  Total ICU stay, i.e, from ICU admission until discharge will be also evaluated at a maximum of 90 days (which is the end of the follow up of the study).

CONTACTS AND LOCATIONS:
Overall Officials: Samir Jaber, MD PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Department of Anesthesiology & Critical Care, St Eloi University Hospital, Montpellier, France

REFERENCES:
- [Derived] Jaber S, Pensier J, Futier E, Paugam-Burtz C, Seguin P, Ferrandiere M, Lasocki S, Pottecher J, Abback PS, Riu B, Belafia F, Constantin JM, Verzilli D, Chanques G, De Jong A, Molinari N; NIVAS Study Group. Noninvasive ventilation on reintubation in patients with obesity and hypoxemic respiratory failure following abdominal surgery: a post hoc analysis of a randomized clinical trial. Intensive Care Med. 2024 Aug;50(8):1265-1274. doi: 10.1007/s00134-024-07522-4. Epub 2024 Jul 29. PMID 39073580
- [Derived] Jaber S, Lescot T, Futier E, Paugam-Burtz C, Seguin P, Ferrandiere M, Lasocki S, Mimoz O, Hengy B, Sannini A, Pottecher J, Abback PS, Riu B, Belafia F, Constantin JM, Masseret E, Beaussier M, Verzilli D, De Jong A, Chanques G, Brochard L, Molinari N; NIVAS Study Group. Effect of Noninvasive Ventilation on Tracheal Reintubation Among Patients With Hypoxemic Respiratory Failure Following Abdominal Surgery: A Randomized Clinical Trial. JAMA. 2016 Apr 5;315(13):1345-53. doi: 10.1001/jama.2016.2706. PMID 26975890